CLINICAL TRIAL: NCT06080698
Title: Gram-Negative Bloodstream Infection Oral Antibiotic Therapy Trial
Acronym: GOAT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00390397; CER-2022C1-26099 (Other Grant/Funding Number: Patient-Centered Outcomes Research Institute (PCORI))
Record Dates: First submitted 2023-10-02; First posted 2023-10-12 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Gram-negative Bacteremia
Keywords: Gram-negative bacteremia; Antibiotic treatment; Antibiotic route; Escherichia coli; Pseudomonas aeruginosa; Klebsiella pneumoniae; Desirability of outcome ranking (DOOR)
MeSH Terms: conditions — Escherichia coli Infections; Pseudomonas Infections | interventions — Anti-Bacterial Agents

STUDY DESIGN:
Intervention Model Description: Eligible participants with GN-BSI will be randomized to (arm 1) IV antibiotics or (arm 2) oral antibiotics for the treatment of GN-BSI.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Intravenous Antibiotics (Active Comparator): IV antibiotics from the time of randomization to the completion of antibiotic treatment. Includes antibiotics such as ceftriaxone, cefepime, piperacillin-tazobactam, and meropenem.
  Interventions: Drug: Intravenous Antibiotics
- Oral Antibiotics (Active Comparator): Oral antibiotics from the time of randomization to the completion of antibiotic treatment, Includes antibiotics such as amoxicillin, cephalexin, ciprofloxacin, and trimethoprim-sulfamethoxazole.
  Interventions: Drug: Oral Antibiotics

INTERVENTIONS:
Drug: Intravenous Antibiotics — Participants will continue to receive intravenous antibiotics until the completion of the treatment course
  Arms: Intravenous Antibiotics
Drug: Oral Antibiotics — Participants will transition to oral antibiotics at the time of randomization and will continue oral antibiotics until the completion of the treatment course
  Arms: Oral Antibiotics

SUMMARY:
The Gram-negative bloodstream infection Oral Antibiotic Therapy trial (The GOAT Trial) is a multi-center, randomized clinical trial that hypothesizes that early transition to oral antibiotic therapy for the treatment of Gram-Negative BloodStream Infection (GN-BSI) is as effective but safer than remaining on intravenous (IV) antibiotic therapy for the duration of treatment.

DETAILED DESCRIPTION:
This is an open-label, pragmatic, randomized trial of approximately 1,204 adult patients hospitalized across 9 United States hospitals with the overarching goal of determining whether the optimal approach for the management of GN-BSI is (1) IV antibiotics for the duration of treatment or (2) initial IV antibiotics followed by early transition to oral antibiotics for the duration of treatment. Patients will be randomized in a 1:1 ratio to remain on IV antibiotics or transition to oral antibiotics as soon as possible after blood culture collection, but no more than 5 days later. The primary objective is to compare the Desirability of Outcomes Ranking (DOOR) distributions between patients with GN-BSI receiving IV antibiotic treatment only versus patients transitioned early to oral antibiotic treatment. The study hypothesis is that oral treatment will result in a more favorable DOOR distribution than IV treatment, likely as a result of differential adverse events and changes in Quality of Life (QoL) profiles.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥ 18 years) at the time of screening
* Hospitalized
* Identification of at least one Gram-negative organism in a blood culture
* Capable of providing written informed consent (includes through a legally authorized representative)
* Willingness to adhere to assigned study arm
* Capable and willing to complete a follow-up QoL interview (including through a legally authorized representative)

Exclusion Criteria:

* Unable to tolerate or absorb a course of oral antibiotics
* Actively receiving vasopressors
* Gram-negative organism not susceptible to any oral antibiotics
* Gram-negative organism not susceptible to any IV antibiotics
* Polymicrobial bloodstream infection

  * The following patients with polymicrobial infections remain eligible for enrollment: (1) more than one morphology or species of a gram-negative organism (except for Acinetobacter baumannii or Stenotrophomonas maltophilia), (2) a single positive blood culture with a common commensal organism (grown in addition to an Enterobacterales species or Pseudomonas aeruginosa
* Allergy or contraindication rendering no oral option or no IV option for therapy with the listed antibiotic agents.
* Anticipated duration of therapy greater than 14 days
* Central nervous system infection
* Absolute neutrophil count of <500 cells/mL or anticipated to reduce to <500 cells/mL during the antibiotic treatment course.
* Receiving hospice care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1204 (Estimated)
Dates: Start 2024-02-22 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Desirability of Outcome Ranking (DOOR) | Day 30
  Each participant will be placed in 1 of 5 DOOR levels based on overall clinical response and treatment-related adverse events (AE). The 5 DOOR levels are as follows: successful clinical response and no treatment-related AE (Level 1); mild suboptimal clinical response or mild treatment-related AE (Level 2); moderate suboptimal clinical response or moderate treatment-related AE (Level 3); significant suboptimal clinical response or significant treatment-related AE (Level 4); death (Level 5). The distribution of participants in the five DOOR levels will be used to ultimately determine which treatment approach is superior for the management of GN-BSI (i.e., IV antibiotic treatment or early transition to oral antibiotic treatment).

SECONDARY OUTCOMES:
Incidence of All Cause Mortality | Day 30
  30-day all cause mortality will be compared between adults with GN-BSI receiving IV antibiotic treatment only versus those transitioned early to oral antibiotic treatment
Frequency of Recurrent infection | Day 30
  30-day recurrent infection with the same bacterial species will be compared between adults with GN-BSI receiving IV antibiotic treatment only versus those transitioned early to oral antibiotic treatment
Length of stay (days) | Day 30
  Hospital length of stay will be compared between adults with GN-BSI alive at day 30 receiving IV antibiotic treatment only versus those transitioned early to oral antibiotic treatment
Number of Participants with Treatment-related adverse events | Day 30
  Moderate to severe treatment-related AEs will be compared between adults with GN-BSI receiving IV antibiotic treatment only versus those transitioned early to oral antibiotic treatment

CONTACTS AND LOCATIONS:
Overall Officials: Pranita D Tamma, MD, MHS, Principal Investigator — Johns Hopkins University; Sara E Cosgrove, MD, MS, Principal Investigator — Johns Hopkins University
Locations (11):
- United States (11):
  - University of California, San Francisco, San Francisco, California
  - Denver Health Hospital Authority, Denver, Colorado
  - University of Maryland Medical Center, Baltimore, Maryland
  - Johns Hopkins University Hospital Systems, Baltimore, Maryland
  - Mayo Clinic, Rochester, Minnesota
  - Rutgers-RWJ University Hospital, New Brunswick, New Jersey
  - Duke University, Durham, North Carolina
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Houston Methodist, Houston, Texas
  - Carilion Clinic, Roanoke, Virginia